CLINICAL TRIAL: NCT05540509
Title: Active Moms: A Feasibility Study of a Community-Based and Home-Based Physical Activity Intervention for Low-Income, Ethnic-Minority Mothers
Brief Title: Active Moms Project: Physical Activity Intervention for Low-Income Mothers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: California State University, Long Beach (Other)
Responsible Party: Principal Investigator, Guido Urizar, Professor, California State University, Long Beach
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PHS 11-252
Record Dates: First submitted 2022-06-28; First posted 2022-09-14 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Physical Inactivity
Keywords: physical activity; community; home; intervention; ethnic minority; mothers
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Intervention Model Description: prospective, convergent mixed-methods, randomized group design
Who Masked: Outcomes Assessor
Masking Description: Staff completing assessments were blind to participants' study condition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Community-based intervention (Experimental): This program consisted of 12 group exercise sessions over a three-month period that were offered in Spanish and English. Each two-hour session consisted of 90 minutes of flexibility, cardiovascular, and strength exercises to meet physical activity recommendations and 30 minutes of group discussions that focused on topics related to the adoption and maintenance of physical activity.
  Interventions: Behavioral: Community-based intervention
- Home-based intervention (Active Comparator): Mothers randomized to the HBI group participated in a three-month program where they were given print-based materials (offered in Spanish or English) at each monthly assessment time point. The print-based materials provided information on multiple cardiovascular, strength training, and flexibility exercises that they could do at home.
  Interventions: Behavioral: Home-based intervention

INTERVENTIONS:
Behavioral: Community-based intervention — Mothers were given physical activity goals and coping resources to practice at home and were asked to record their experiences on an activity log. Course content was taught from a detailed training manual and was based on concepts and strategies from social cognitive theory that have been effective in increasing physical activity and fitness levels among mothers. In the first month, mothers attended group exercise sessions twice per week (total of eight group sessions) and exercised on their own once per week. In the second month, mothers attended group exercise sessions once per week (total of four group sessions) and exercised on their own twice per week. In the third month, mothers exercised on their own three times per week.
  Other Names: CBI
  Arms: Community-based intervention
Behavioral: Home-based intervention — The HBI group received information on building social support and reducing physical activity barriers based on materials from the Diabetes Prevention Program. Participants were also given activity logs to record their physical activity each week, which was collected by research staff at each monthly assessment time point to assess how participants were progressing with their physical activity goals. Mothers exercised on their own for three months with the goal of meeting national physical activity guidelines
  Other Names: HBI
  Arms: Home-based intervention

SUMMARY:
Despite the health benefits of physical activity, increasing regular physical activity levels among low-income, ethnic-minority mothers has remained a significant challenge. The current mixed-methods feasibility study explored the impact that a three-month community-based (CBI) and a home-based intervention (HBI) had on improving physical activity and fitness levels, as well as psychosocial outcomes (self-efficacy and social support) among low-income, ethnic-minority mothers. These results support the efficacy of CBIs and HBIs in improving PA and fitness levels and have important implications for improving health outcomes among low-income, ethnic-minority mothers.

DETAILED DESCRIPTION:
Despite the health benefits of physical activity, increasing regular physical activity levels among low-income, ethnic-minority mothers has remained a significant challenge. Yet, few studies have examined the feasibility of implementing interventions to address physical activity barriers often experienced by this population. The current mixed-methods feasibility study explored the impact that a three-month community-based (CBI) and a home-based intervention (HBI) had on improving physical activity and fitness levels, as well as psychosocial outcomes (self-efficacy and social support) among low-income, ethnic-minority mothers. Thirty mothers were randomized to either a three-month community-based intervention (CBI) or a home-based intervention (HBI) and completed pre- and post-intervention assessments of physical activity (self-report, accelerometer), fitness (cardiorespiratory, muscle endurance and strength, flexibility), self-efficacy, and social support. Post-intervention focus groups were also conducted. Through formative research, this pilot work will develop and empirically test a CBI and HBI among low-income mothers for use in local community centers. The results of the proposed work have substantial public health implications and are expected to advance the investigator's understanding of how low-income mothers effectively use these intervention modalities to adopt healthy behaviors and produce change that can positively impact their health, as well as that of their children. Further, the proposed research will yield two physical activity interventions that can be readily delivered in community settings, are scalable, and are relatively low cost. Finally, these results will help identify those subgroups of mothers that may do particularly well (or poorly) with these innovative approaches to physical activity adoption and maintenance. This has important implications for the tailoring of physical activity programs to individual needs and preferences.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* a mother of a young child (<10 years of age)
* fluent in either Spanish or English
* Sedentary (i.e., not engaging in 90 minutes or more of moderate or vigorous physical activity per week)

Exclusion Criteria:

* Not medically cleared by a doctor or by a medical history screener to engage in moderate-intensity physical activity
* Currently pregnant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-05-23 (Actual); Primary Completion 2013-05-01 (Actual); Study Completion 2013-05-01 (Actual)

PRIMARY OUTCOMES:
Change in Physical Activity from baseline to 3 months post-intervention | Self-reported and fitbit physical activity assessments were conducted at baseline and at one, two, and three months post-intervention.
  Self-reported duration of moderate/vigorous physical activity was assessed using the Check and Line Questionnaire (CALQ), with higher numbers representing greater average minutes of moderate/vigorous-intensity PA completed/day over a three-day assessment period. Objective physical activity was assessed using the Fitbit One (2009 version), which is an accelerometer worn on the hip (clipped to a participant's clothing at the waist). For the current study, very active minutes were examined (measure of basal metabolic rate/minute). Activity data was averaged across the three days that the Fitbit was worn, with greater number of very active minutes indicating greater daily moderate/vigorous-intensity physical activity levels.
Change in Cardiorespiratory Fitness from baseline to 3 months post-intervention | Cardiorespiratory fitness assessments were conducted at baseline and at one, two, and three months post-intervention.
  Cardiorespiratory fitness was assessed via predicted relative maximum oxygen consumption, also known as relative VO2 max (ml/kg/min) after participants completed a timed mile walk, with a greater relative VO2 max being an indicator of greater cardiorespiratory fitness.
Change in Muscle Endurance from baseline to 3 months post-intervention | Muscle endurance assessments were conducted at baseline and at one, two, and three months post-intervention.
  Muscle endurance was assessed by the number of modified push-ups completed in correct form, with a greater number of 90° push-ups completed representing greater muscular endurance.
Change in Flexibility from baseline to 3 months post-intervention | Flexibility assessments were conducted at baseline and at one, two, and three months post-intervention.
  Flexibility was assessed by a modified sit and reach test (in inches) where mothers were instructed to reach forward as far as they could with their hands over each other, over a three-foot ruler, without removing their body from the wall and holding this position for at least two seconds, with greater inches indicating greater flexibility.

SECONDARY OUTCOMES:
Change in Physical Activity Self-Efficacy from baseline to 3 months post-intervention | Physical Activity Self-efficacy assessments were conducted at baseline and at one, two, and three months post-intervention.
  Physical Activity Self-efficacy was assessed using the Barriers Self-Efficacy Scale. The 14-item Barriers Self-Efficacy Scale measures a mother's level of confidence in engaging in physical activity despite barriers experienced over the next three months, with higher scores (range=0-100) reflecting higher self-efficacy for physical activity in the face of barriers.
Change in Fitness Self-Efficacy from baseline to 3 months post-intervention | Fitness Self-efficacy assessments were conducted at baseline and at one, two, and three months post-intervention.
  Fitness Self-efficacy was assessed using the Self-Efficacy for Physical Performance Scale. The 5-item Self-Efficacy for Physical Performance Scale measures a participant's self-efficacy to currently perform multiple activities that improve fitness (e.g., walking a mile, doing push-ups), with higher scores (range=0-100) indicating higher self-efficacy for fitness.
Change in Social Support from baseline to 3 months post-intervention | Social support assessments were conducted at baseline and at one, two, and three months post-intervention.
  Social support for physical activity was assessed using the 15-item Social Support for Exercise Survey. The Social Support for Exercise Survey measures the degree of social support received from one's family and friends to engage in physical activity, with higher scores (range=0-75) reflecting more social support received from each of these support networks.

CONTACTS AND LOCATIONS:
Overall Officials: Guido Urizar, PhD, Principal Investigator — California State University, Long Beach

IPD SHARING:
Plan to Share IPD: No
Due to the sensitive nature of the questions asked in this study, survey respondents were assured raw data would remain confidential and would not be shared.
  Data not available / The data that has been used is confidential